CLINICAL TRIAL: NCT04234061
Title: A Phase II, Open-Label, Single Arm Trial to Assess The Efficacy and Safety of the Combination of Tisagenlecleucel And Ibrutinib in Mantle Cell Lymphoma
Brief Title: Clinical Trial to Assess The Efficacy and Safety of the Combination of Tisagenlecleucel And Ibrutinib in Mantle Cell Lymphoma
Acronym: TARMAC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19/008
Record Dates: First submitted 2020-01-05; First posted 2020-01-21 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Mantle Cell Lymphoma Recurrent
Keywords: ibrutinib; Tisagenlecleucel; Chimeric Antigen Receptor - Tcell (CAR-T); B-cell non-Hodgkin lymphoma; TP53 mutation; bruton's tyrosine kinase (BTK) inhibitor
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — ibrutinib; tisagenlecleucel

STUDY DESIGN:
Intervention Model Description: single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single (Experimental): ibrutinib and Tisagenlecleucel
  Interventions: Combination Product: ibrutinib and Tisagenlecleucel

INTERVENTIONS:
Combination Product: ibrutinib and Tisagenlecleucel — Single-arm study investigating combination of ibrutinib and Tisagenlecleucel treatment

SUMMARY:
This is an open label, multi-center, single-arm, phase II study investigating the efficacy and safety of the combination of ibrutinib and Tisagenlecleucel in twenty patients with relapsed or refractory Mantle Cell Lymphoma (MCL) or who had sub-optimal response to standard therapy in the presence of TP53 mutation.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all the following criteria for study entry:

  1. Written informed consent prior to screening procedures
  2. Be ≥18 years of age on the day of signing informed consent
  3. Have a confirmed diagnosis of MCL according to World Health Organization (2016) criteria
  4. Have sufficient fresh or archival material available for central review
  5. At least one site of radiographically assessable disease not previously irradiated (lymph node with largest diameter ≥1.5cm, or unequivocal evaluable hepatomegaly/splenomegaly or marrow phase disease)
  6. Meet at least one of the following disease criteria:

     * Have relapsed, or progressed following at least 1 prior line of systemic chemoimmunotherapy for MCL (may include ibrutinib or other BTK-inhibitor in combination)
     * Be refractory to at least one prior line of chemoimmunotherapy (refractory is defined as less than a conventional PR following 2 cycles of anthracycline or cytarabine-containing therapy)
     * Have achieved <CR on PET imaging following 2 cycles of anthracycline or cytarabine-containing therapy in the presence of aberrations of p53; or <CR post autologous stem cell transplantation
     * Failure to achieve CR following at least 6 months of an ibrutinib or BTK inhibitor -containing front-line regimen, or failure to achieve PR following 8 weeks of a BTK inhibitor
  7. Have a life expectancy of ≥ 3 months, as judged by the investigator
  8. Have acceptable haematological function within 7 days prior to registration, defined as:

     * Absolute neutrophil count ≥1x10^9/L (may be supported by growth)
     * Absolute lymphocyte count ≥0.3x10^9/L or absolute CD3+ fraction > 0.15x 10^9/L
     * Platelets >50x 10^9/L unless explained by lymphoma at the discretion of the CPI
     * Haemoglobin ≥ 80 g/L (may be transfusion supported)
  9. Have acceptable organ function within 7 days prior to registration, defined as:

     * Serum creatinine ≤1.5 x ULN, or a calculated creatinine clearance of at least 50 mL/min using the Cockcroft-Gault equation (see appendix 1) or a 24-hour urine collection
     * AST or ALT ≤3.0 x ULN
     * Bilirubin ≤ 1.5 x ULN (with the exception of patients with Gilbert's syndrome. Patients with Gilbert's syndrome may be included if their total bilirubin is ≤3.0 x ULN and direct bilirubin ≤1.5 x ULN).
     * aPTT and PT ≤ 1.5x ULN
     * Adequate pulmonary function defined as:
* No or mild dyspnea (≤ grade 1)
* Oxygen saturation measured by pulse oximetry ≥ 90 percent on room air 10. Female patients of childbearing potential and non-sterile male patients (with partners of childbearing potential) must agree to use highly effective methods of contraception from registration on the study to 30 days after the last dose of ibrutinib and 12 months after Tisagenlecleucel infusion and until Tisagenlecleucel is no longer present by qPCR on two consecutive tests (whichever is later):

  * Total abstinence from sexual intercourse when this is in line with the preferred and usual life style of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Female sterilisation (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or bilateral tubal ligation at least six weeks prior to registration. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment
  * Male sterilisation (at least 6 months prior to screening). For female patients on the study, the vasectomised male partner should be the sole partner for that patient
  * Use of oral, (estrogen and progesterone), injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception. In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before enrolment into this study.

Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment is she considered not of child bearing potential.

11. Female patients of childbearing potential must have a negative serum (beta-human chorionic gonadotropin (β-hCG) or urine pregnancy test within 7 days of registration 12. Sexually active male patients must use a condom during intercourse and must agree to refrain from sperm donation, from registration on the study until 30 days after the last dose of ibrutinib or 12 months after Tisagenlecleucel infusion and until Tisagenlecleucel is no longer present by qPCR on two consecutive tests

Exclusion Criteria:

* Patients who meet any of the following criteria will be excluded from study entry:

  1. Prior allogeneic transplantation
  2. Autologous transplantation within 6 weeks prior to registration
  3. Active and uncontrolled autoimmune cytopenias
  4. Active central nervous system involvement with MCL
  5. Previous treatment with adoptive T-cell therapy
  6. Receipt of a non BTK-inhibitor investigational medical product within the last 30 days prior to planned leukapheresis
  7. Receipt of a non-anti CD20- monoclonal antibody with anti-neoplastic intent within 30 days prior to planned leukapheresis
  8. Receipt of steroids >20mg prednisolone or equivalent in the fortnight prior to planned leukapheresis
  9. Requirement for ongoing therapy with:

     * Potent CYP3A inhibitors (e.g. indinavir, ketoconazole, clarithromycin)
     * Potent CYP3A inducers (e.g. rifampin, phenytoin, carbamazepine)
     * Vitamin K antagonists (e.g. warfarin or equivalent)
     * Antiretroviral medications
  10. Consumption within 3 days prior to registration:

      * Grapefruit or grapefruit products
      * Seville oranges
      * Star fruit
  11. Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure or myocardial infarction within 6 months of screening or class III to IV cardiac disease as defined by the New York Heart Association Functional Classification
  12. Active neurological disorders of clinical relevance (e.g. epilepsy, severe brain injury, dementia, Parkinson's disease or autoimmune/inflammatory disorders (e.g. Guillain-Barre syndrome, motor neurone disease, chronic inflammatory demyelinating polyneuropathy)
  13. Other significant life-threatening illness or medical condition which, in the investigator's opinion, could compromise the subject's safety, interfere with absorption or metabolism of study drug, or put the study outcomes at undue risk
  14. History of other active malignancy, with the exception of:

      * Adequately treated in situ carcinoma of the cervix or breast
      * Adequately treated basal cell carcinoma of skin or localised squamous cell carcinoma of the skin
      * Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent and without evidence of recurrence for at least 2 years prior to registration
  15. History of human immunodeficiency (HIV) or active hepatitis C virus or active hepatitis B virus. NOTE: Serology must be repeated at the pre-conditioning stage prior to infusion with Tisagenlecleucel.
  16. Clinically significant active infection confirmed by clinical evidence, imaging or positive laboratory tests (e.g. blood cultures, viral DNA/RNA by PCR)
  17. Receipt of live, attenuated vaccines within 4 weeks of registration
  18. Major surgery within 4 weeks prior to registration
  19. Pregnant or nursing (lactating) women. Note: Women of child-bearing potential must have a negative serum pregnancy test performed within 24 hours before leukapheresis, lymphodepletion (if performed) and prior to Tisagenlecleucel infusion.
  20. Known hypersensitivity to the excipients of Tisagenlecleucel or to any product to be given to the patient as per the study protocol (e.g. tocilizumab and lymphodepleting agents)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Estimate complete response (CR) rate at month 4 following the infusion of Tisagenlecleucel using the Lugano criteria | 4 months after Tisagenlecleucel infusion using the Lugano criteria
  Using the Lugano criteria

SECONDARY OUTCOMES:
Evaluate safety of combination therapy with Tisagenlecleucel and ibrutinib through monitoring of the incidence, nature and severity of adverse events (graded according to NCI CTCAE v5.0), SAEs, dose interruptions and dose reductions of ibrutinib | From date of registration until the date of first progression or until the date of death from any cause, whichever occurs first, assessed up to the date of the patient's last annual assessment, on average for five years
  Through monitoring of the incidence, nature and severity of adverse events (graded according to NCI CTCAE v5.0), Serious Adverse Events, dose interruptions and dose reductions of ibrutinib
Estimate objective response (OR) rate at day 28, month 4, 6, 9 and 12 following the infusion of Tisagenlecleucel using Lugano criteria | day 28, month 4, 6, 9 and 12 following the infusion of Tisagenlecleucel
  Using Lugano criteria
To estimate objective response (OR) rate at day 28, month 4, 6, 9 and 12 following the infusion of Tisagenlecleucel by TP53 status | day 28, month 4, 6, 9 and 12 following the infusion of Tisagenlecleucel by TP53 status
  Assessment of TP53 status
To estimate Minimal Residual Disease (MRD) negative response rates by aggregate measure of peripheral blood/or bone marrow flow cytometry, PCR and ctDNA | At day 28, months 4, 6, 9 and 12 following the infusion of Tisagenlecleucel
  Measured through aggregate measure of peripheral blood/or bone marrow flow cytometry, PCR and ctDNA
To estimate progression-free survival | From date of registration until the date of first progression or until the date of death from any cause, whichever occurs first, assessed up to the date of the patient's last annual assessment, on average for five years
  According to Lugano criteria
To estimate duration of response | From date of registration until the date of first progression or until the date of death from any cause, whichever occurs first, assessed up to the date of the patient's last annual assessment, on average for five years
  Using Lugano criteria
To estimate overall survival | From date of registration until the date of first progression or until the date of death from any cause, whichever occurs first, assessed up to the date of the patient's last annual assessment, on average for five years
  By monitoring for patient death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dickinson, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter Mac Callum Cancer Centre, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Minson A, Hamad N, Cheah CY, Tam C, Blombery P, Westerman D, Ritchie D, Morgan H, Holzwart N, Lade S, Anderson MA, Khot A, Seymour JF, Robertson M, Caldwell I, Ryland G, Saghebi J, Sabahi Z, Xie J, Koldej R, Dickinson M. CAR T cells and time-limited ibrutinib as treatment for relapsed/refractory mantle cell lymphoma: the phase 2 TARMAC study. Blood. 2024 Feb 22;143(8):673-684. doi: 10.1182/blood.2023021306. PMID 37883795